CLINICAL TRIAL: NCT04273425
Title: Bone Pain in Multiple Myeloma- a Translational Study
Acronym: BPMM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: STH20993
Record Dates: First submitted 2020-02-06; First posted 2020-02-18 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma
Keywords: Pain
MeSH Terms: conditions — Multiple Myeloma; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Myeloma cells will be collected and frozen for subsequent genetic analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study cohort (Confirmed myeloma patients): Patients with suspected multiple myeloma will be recruited. They will be asked to fill in questionnaires (regarding pain, quality of life, catastrophizing), donate serum samples and allow the research team to access their clinical data and their diagnostic bone biopsy.
  Those who receive a positive diagnosis will be followed up upon completion of first-line treatment, and questionnaire data and blood samples collected again.
- Control cohort (non-confirmed myeloma patients): Patients with suspected multiple myeloma will be recruited. They will be asked to fill in questionnaires (regarding pain, quality of life, catastrophizing), donate serum samples and allow the research team to access their clinical data and their diagnostic bone biopsy.
  Samples from patients who receive a negative myeloma diagnosis will be used as negative controls.

SUMMARY:
While the survival expectancy of myeloma patients continues increasing due to the discovery of novel treatments, bone pain remains one of the main symptoms of this patient population, impairing their mood and quality of life.

The aim of this study is to characterize the subjective experience of pain in myeloma patients, and its correlation with disturbances in serum biomarkers and bone innervation.

Primary research questions:

How is the bone pain experienced by myeloma patients (intensity, location and type of pain) and how does it affect their quality of life?

Do myeloma cells induce changes in the density and/or location of nerve fibres innervating the bone, and if so, are these correlated to the pain experience?

Secondary research questions:

Are the alterations in the bone innervation of myeloma patients similar to those of immunocompetent animal models of the disease (the 5TGM1 model)?

Is serum paraprotein correlated with the subjective experience of myeloma-induced bone pain?

Are the bone turnover biomarkers (C-terminal telopeptides Type 1 collagen, CTX, and procollagen type 1 N-terminal propeptide, P1NP) and inflammatory serum biomarkers correlated with the subjective experience of myeloma-induced bone pain?

Do myeloma cells affect the location, number or density of bone cells (e.g. osteoblasts, osteoclasts)?

DETAILED DESCRIPTION:
Patients undergoing diagnostic procedures (i.e. trephine bone biopsy) for suspected multiple myeloma will be invited to participate in the study, and provided with time to consider their participation.

Patients who consent will be provided with a set of seven standardized questionnaires assessing their pain, quality of life and catastrophizing. Additionally, patients will be asked to fill in demographic information.

Consenting patients will be asked to donate a fasting blood sample and give permission to the research team to retrieve their triphane bone biopsy, once the medical team has finished evaluating it. The presence, location and density of nerve fibres innervating the bone will be evaluated. Patients will also be consented to allow retrieval of medical information from their medical records, and correlations between serum biomarkers, disturbances in bone innervation, paraprotein levels, etc. and their self-reported experience of pain will be investigated. Patients with a negative diagnosis for multiple myeloma (expectably monoclonal gammopathy of undetermined significance (MGUS) patients) will be used as negative controls.

Patients who receive a positive diagnosis for multiple myeloma will be asked to fill in the same set of questionnaires upon completion of the first-line treatment (approximately 7 to 8 months after baseline assessment). Fasting serum blood samples will be collected. To evaluate treatment´s success, it is common medical practice to extract a new trephine bone biopsy upon completion of first line treatment. The research team will access these biopsies and evaluate the presence, density and location of nerve fibres in bone. Changes in nerve fibre profiles, serum biomarkers and the self-reported experience of pain, quality of life and catastrophizing following first-line treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Undergoing diagnostic procedures for suspected myeloma (no previous treatment for this)
* Patients who are local to Sheffield (or who are local to any other institute that may join in collaboration)
* Must be able to give informed consent

Exclusion Criteria:

* Patient who are unable to give consent
* Patients who do not speak English
* Patients who are too unwell to be recruited
* Patients who have had recent chemotherapy for different malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing diagnostic procedures for suspected multiple myeloma at Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield, UK.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in bone innervation by immunohistological assessment (presence) | Change from baseline to completion of first line treatment (expected to be measured at 8 months after baseline; expected to be reported within 2 years from baseline) for patients with a positive myeloma diagnosis.
  The presence of sympathetic and sensory nerve fibers innervating the bone will be assessed in the diagnostic trephine bone biopsies.
Change in bone innervation by immunohistological assessment (location) | Change from baseline to completion of first line treatment (expected to be measured at 8 months after baseline; expected to be reported within 2 years from baseline) for patients with a positive myeloma diagnosis.
  The location sympathetic and sensory nerve fibers innervating the bone will be assessed in the diagnostic trephine bone biopsies.
Change in bone innervation by immunohistological assessment (density) | Change from baseline to completion of first line treatment (expected to be measured at 8 months after baseline; expected to be reported within 2 years from baseline) for patients with a positive myeloma diagnosis.
  The density of sympathetic and sensory nerve fibers innervating the bone will be assessed in the diagnostic trephine bone biopsies.
Characterization of pain in patients with firstly-diagnosed myeloma through standardized questionnaires (Brief Pain Inventory (BPI), FACT-BP(FACT-Bone Pain), PCS (Pain catastrophizing scale), painDETECT) | Baseline
  Questionnaires will be used to characterize the self-reported experience of pain in patients with firstly-diagnosed myeloma
Characterization of quality of life in patients with firstly-diagnosed myeloma through standardized questionnaires (EORTC QLQ-C30 (core 30) , EORT QLQ-MY20 (myeloma module 20), EORTC QLQ-CIPN20 (chemotherapy-induced peripheral neuropathy module 20) ) | Baseline
  Questionnaires will be used to characterize the quality of life of patients with firstly-diagnosed myeloma
Change in quality of life in myeloma after first-line treatment through standardized questionnaires (EORTC QLQ-C30, EORT QLQ-MY20, EORTC QLQ-CIPN20) | Change from baseline to completion of first line treatment (expected to be measured at 8 months after baseline; expected to be reported within 2 years from baseline) for patients with a positive myeloma diagnosis.
  Questionnaires will be used to characterize the quality of life of patients with firstly-diagnosed myeloma and after completion of first-line treatment
Change in pain in myeloma after first-line treatment through standardized questionnaires (BPI, FACT-BP, PCS, painDETECT) | Change from baseline to completion of first line treatment (expected to be measured at 8 months after baseline; expected to be reported within 2 years from baseline) for patients with a positive myeloma diagnosis.
  Questionnaires will be used to characterize the experience of pain in patients with firstly-diagnosed myeloma and after completion of first-line treatment

SECONDARY OUTCOMES:
Change in serum bone biomarkers (CTX1, P1NP) measured by ELISA | Change from baseline to completion of first line treatment (expected to be measured at 8 months after baseline; expected to be reported within 2 years from baseline) for patients with a positive myeloma diagnosis.
  Measurement of bone turnover biomarkers in serum samples through enzyme-linked immunosorbent assay (ELISA).
Change in inflammatory serum biomarkers measured by multiplex array. | Change from baseline to completion of first line treatment (expected to be measured at 8 months after baseline; expected to be reported within 2 years from baseline) for patients with a positive myeloma diagnosis.
  Measurement of an set of inflammatory cytokines in serum samples through multiplex cytokine arrays.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Chantry, MD, PhD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be collected, stored and analyzed. The results of the study will be published in peer-reviewed scientific journals. Individual participant data will not be shared with the scientific or medical community unless specifically requested.

REFERENCES:
- [Derived] Diaz-delCastillo M, Andrews RE, Mandal A, Andersen TL, Chantry AD, Heegaard AM. Bone Pain in Multiple Myeloma (BPMM)-A Protocol for a Prospective, Longitudinal, Observational Study. Cancers (Basel). 2021 Mar 30;13(7):1596. doi: 10.3390/cancers13071596. PMID 33808348